CLINICAL TRIAL: NCT00314756
Title: Topical Imiquimod 5% Cream in the Treatment of Nodular Basal Cell Carcinoma After Initial Treatment With Curettage
Brief Title: Treatment of Nodular Basal Cell Carcinoma (BCC) With Imiquimod 5% Cream After Curettage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG04-484
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2005-03

CONDITIONS: Basal Cell Carcinoma
Keywords: imiquimod cream; nodular basal cell carcinoma; curettage
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Imiquimod

INTERVENTIONS:
Drug: imiquimod

SUMMARY:
To assess the efficacy of treating a nodular basal cell carcinoma with imiquimod cream after initial treatment with curettage

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of imiquimod 5% cream on nodular BCC lesions treated 5x/week for 6 weeks after primary treatment with curettage without electrodesiccation. The secondary objective of this study is to evaluate the cosmetic outcome after treatment of the lesions using this modality.

ELIGIBILITY:
Inclusion Criteria:

1. Are willing and able to give informed consent;
2. Are at least 18 years of age;
3. Are willing to comply with all study requirements, evaluations, and procedures
4. Have 1 clinically typical, visible nodular BCC lesion which meets the following criteria:

   * a primary lesion (not recurrent, not previously treated or biopsied)
   * non-infected
   * size between 0.25 and 1.5 cm2
   * located at least 1 cm from the eyes, nose, mouth, ear, and hairline to exclude the H-zone of the face
   * clinically consistent with nodular BCC
   * histologically consistent with nodular BCC and have no histological evidence of a morpheaform or micronodular pattern
   * suitable for treatment with surgical excision
   * easily identifiable and treatable by subject or reliable subject representative
5. Are free of any significant physical abnormalities or previous scarring in the potential application site area that may cause difficulty with examinations.
6. Are willing to stop using over-the-counter retinol products or products containing alpha or beta hydroxyacids in the treatment and surrounding area 8 hours prior to treatment with the imiquimod cream and clinic visits.

Exclusion Criteria:

1. Have evidence of clinically significant, unstable, cardiovascular or immunosuppressive, hematologic, hepatic, neurologic, renal, endocrine, collagen-vascular, or gastrointestinal abnormalities or disease that may interfere with completion of the study.
2. Have any dermatological disease in the treatment or surrounding area that may be exacerbated by treatment with imiquimod or cause difficulty with examination.
3. Have a BCC lesion located within 1 cm of the eyes, nose, mouth, ear, and hairline.
4. Are pregnant at the screening or treatment initiation visit.
5. Have known allergies to any excipient in the study cream
6. Have undergone any surgical procedures in the potential treatment area within 4 weeks of the screening/treatment initiation visit. In addition, skin in the potential application area must be healed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2005-03; Study Completion 2005-11

PRIMARY OUTCOMES:
histologic clearance of basal cell carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Phillip M Williford, MD, Principal Investigator — Wake Forest University Medical Center
Locations (1):
- Wake Forest University Medical Center, Winston-Salem, North Carolina, United States